CLINICAL TRIAL: NCT03727776
Title: Adrenocorticotropic Hormone for Intraocular Inflammation in Post-operative Proliferative Vitreoretinopathy Patients
Brief Title: Adrenocorticotropic Hormone (ACTH) for Post-op Inflammation in Proliferative Vitreoretinopathy (PVR)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00179012
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: Post-operative Intraocular Inflammation
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- H.P. Acthar ® (Experimental): Subjects will self-administer subcutaneous injections of 80 units of adrenocorticotropic hormone analog starting on post-operative day 1 for twice a week until week 8.
  Interventions: Drug: Adrenocorticotropic Hormone
- Controls (No Intervention): Subjects will be managed per the standard of care.

INTERVENTIONS:
Drug: Adrenocorticotropic Hormone — Adrenocorticotropic hormone (ACTH) is a melanocortin peptide hormone that is normally produced in the pituitary gland and acts as a major regulator of adrenal cortex function. It stimulates the adrenal cortex to produce and secrete glucocorticoids. ACTH is available for clinical usage as an injectable gel (H.P. Acthar®).
  Other Names: H.P. Acthar Gel; Repository Corticotropin Injection
  Arms: H.P. Acthar ®

SUMMARY:
This is a pilot study to measure levels of albumin and inflammatory cytokines [including Transforming Growth Factor-Beta (TGF-β) and Interleukin-1 Beta (IL-1β)] in the aqueous humor of post-operative proliferative vitreoretinopathy patients receiving subcutaneous injections of H.P. Acthar®, an adrenocorticotropic hormone (ACTH) analog. The study will be conducted at the Wilmer Eye Institute, Johns Hopkins Hospital. A total of 15 patients will be enrolled and randomized 2:1 to H.P. Acthar® or standard of care. Treatment duration will be 8 weeks and study duration will be 12 weeks. There will be a total of 7 study visits (baseline, day of surgery, post-operative day 1, week 1, week 4, week 8, and week 12).

Subjects will self-administer subcutaneous injections of 80 units of H.P. Acthar® starting on post-operative day 1 for twice a week until week 8. Subjects in the control arm will be managed per the standard of care. Aqueous samples will be obtained at the onset of surgery, 1 day, 1 week and 8 weeks after surgery. Aqueous levels of albumin and inflammatory cytokines (including TGF-β and IL-1β) will be measured at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent and authorization of use and disclosure of protected health information
* Patients undergoing surgery for retinal detachment due to PVR

Exclusion Criteria:

* Patients with poorly controlled diabetes mellitus (defined as HbA1C ≥ 8.0% on any anti-diabetic medications or insulin. If the patient is using any anti-diabetic medication/insulin, he becomes eligible if the medication is used continuously for >30 days)
* Patients with poorly controlled hypertension (defined as systolic blood pressure >180 mm Hg and/or diastolic blood pressure >100 mm Hg at rest with up to 3 anti-hypertensive medications. If a patient's initial measurement exceeds these values, a second reading may be taken 30 or more mins later. If the patient is using any anti-hypertensives, he becomes eligible if the medication is used continuously for >30 days)
* Patients with congestive heart failure
* Patients with scleroderma
* Patients with osteoporosis
* Patients with active systemic fungal infection
* Patients with active ocular herpes simplex
* Patients with prior or active bleeding peptic ulcer
* Pregnant patients or patients who wish to become pregnant during the course of the study (females of child-bearing age will be counselled to use contraception for the duration of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Change in mean aqueous levels of albumin in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 day after surgery, 8 weeks after surgery
  The levels of albumin in the aqueous humor are indicative of blood-retinal barrier breakdown and will be measured in mg/dl
Change in mean aqueous levels of TGF-B in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 day after surgery, 8 weeks after surgery
  The levels of TGF-B in the aqueous humor are indicative of intraocular inflammation and will be measured in mg/dl
Change in mean aqueous levels of interleukin-1B (IL-1B) in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 day after surgery, 8 weeks after surgery
  The levels of IL-1B in the aqueous humor are indicative of intraocular inflammation and will be measured in mg/dl

SECONDARY OUTCOMES:
Change in mean aqueous levels of albumin in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 day after surgery, 1 week after surgery
  The levels of albumin in the aqueous humor are indicative of blood-retinal barrier breakdown and will be measured in mg/dl
Change in mean aqueous levels of TGF-B in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 day after surgery, 1 week after surgery
  The levels of TGF-B in the aqueous humor are indicative of intraocular inflammation and will be measured in mg/dl
Change in mean aqueous levels of interleukin-1B (IL-1B) in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 day after surgery, 1 week after surgery
  The levels of IL-1B in the aqueous humor are indicative of intraocular inflammation and will be measured in mg/dl
Change in mean grade of aqueous cell in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | 1 week, 4 weeks, 8 weeks and 12 weeks after surgery
  Aqueous cell is a clinical indicator of blood-retinal barrier breakdown and intraocular inflammation. It is assessed on slit-lamp examination and is graded on a scale from 0 to 4+, with 0 meaning no aqueous cell and 4+ meaning severe aqueous cell
Change in mean grade of flare in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | 1 week, 4 weeks, 8 weeks and 12 weeks after surgery
  Flare is a clinical indicator of blood-retinal barrier breakdown and intraocular inflammation. It is assessed on slit-lamp examination and is graded on a scale from 0 to 4+ with 0 meaning no flare and 4+ means severe flare
Change in best-corrected visual acuity as measured by Early Treatment of Diabetic Retinopathy Study (ETDRS) score in post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls | Baseline, 1 week, 4 weeks, 8 weeks and 12 weeks after surgery
  The ETDRS score is a standardized score to assess visual acuity used in clinical research. The score ranges from 0 to 100, with higher scores corresponding to better visual acuity (a score of 100 corresponding to a Snellen visual acuity of 20/10).
Percentage of post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls who develop recurrent retinal detachment | 12 weeks after surgery
  Recurrent retinal detachment is a common complication of PVR. It will be diagnosed based on clinical exam and supporting information from diagnostic tests such as Optical Coherence Tomography.
Percentage of post-operative PVR patients receiving subcutaneous injections of H.P. Acthar® versus controls who develop macular edema | 12 weeks after surgery
  Macular edema is a common complication of intraocular surgery. It will be diagnosed based on clinical exam and supporting information from diagnostic tests such as Optical Coherence Tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Wilmer Eye Institute, Johns Hopkins School of Medicine
Locations (1):
- Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore, Maryland, United States